CLINICAL TRIAL: NCT04206566
Title: PHASTER - Pre-Hospital Advanced Airway Management STudying Expedited Routines
Brief Title: Pre-hospital Advanced Airway Management Studying Expedited Routines
Acronym: PHASTER
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Mikael Gellerfors, Head of Research & Development, Swedish Air Ambulance (SLA), Karolinska Institutet
Other Study IDs: PHASTER-01
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Emergency Medicine; Airway Management; Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the Scandinavian and Swiss HEMS critical care teams, the prehospital tracheal intubations (TI) are performed by airway experts with high success rates and low rates of complications. Due to environmental conditions these are today frequently performed in-cabin before take-off. There are so far no published data on comparing outside and in-cabin TI under these circumstances.

This will therefore be the first prospective study comparing prehospital TIs outside or incabin, performed by airway experts.

DETAILED DESCRIPTION:
Background Seriously ill or injured patients might require prehospital TI, which is a potentially lifesaving intervention. Performing TI in a prehospital context differ from the preconditions inhospital due to environmental and technical aspects and resources available (3). Today there is a consensus that prehospital critical care should at least be on the same standards as in-hospital care. The trend therefore has been towards more rigorous safety precautions introducing Standard Operating Procedures (SOP) including 360oaccess to patients with all equipment at close hand brought out from the helicopter or the ambulance and long challenge-response lists. This will shift focus towards adherence to SOPs instead of tailoring the sequence of procedures according to circumstances and patient needs. An experienced operator can plan and communicate appropriate actions from a risk-benefit perspective in a stressful situation. Prehospital interventions have to be time effective, especially where short on-scene times are preferable in time-critical conditions such as uncontrolled internal haemorrhage and traumatic brain injuries.

A recent Nordic multicentre study, PHAST, shows that emergency systems staffed with highly experienced anaesthetists can perform prehospital TI with high success rates, low incidence of complications and short on-scene times. Due to environmental factors, weather and light conditions in the Scandinavian countries, it is not always favourable to perform TI outside the helicopter or ambulance, with 360o -access. Technical aspects in-helicopter/in-ambulance such as access to better suctioning and stretcher positioning, can influence the operator's decision on where to perform the TI. Whether the location of the TI affects the outcome has not yet been studied. A recent experimental mannequin study, SPRINT, suggests that in-cabin intubations can offer equal to, or even better conditions than out of cabin and can shorten on-scene time. To investigate whether this applies to real life conditions, a prospective large-scale clinical study must be done.

Performing prehospital TI is dependent on a well-functioning team where the operator has an assistant backing up during the procedures. The assistants' level of airway experience and the teams' accumulated experience working together has not been studied earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of prehospital drug-assisted intubation.

Exclusion Criteria:

* All cases where prehospital TI is performed without the use of any drugs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All drug-assisted intubations performed at the participating HEMSorganizations between 01/01/2020 and 01/09/2021.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
First pass success rate on prehospital tracheal intubation | While handling the patient in need for tracheal intubation
  Successful intubation is defined as the endotracheal tube verified in the trachea. Prehospital intubations are performed outside the hospitals by ambulance helicopter personnel.

SECONDARY OUTCOMES:
Tracheal intubation performed outside or in-cabin (in helicopter or in ambulance) | While handling the patient case
  The location of the procedure
Number of tracheal intubation attempts | While handling the patient case
Perceived difficulty of tracheal intubation | While handling the patient case
  Measured on a numeric analogue scale
Time to perform tracheal intubation | While handling the patient case
  Time from first passing teeth with laryngoscope to tube verification with ETCO2 and lung auscultation.
Complications related to the drug assisted intubation | While handling the patient case
Prehospital mortality | While handling the patient case
Scene time 1 | While handling the patient case
  Measured from entering patient zone (<3 m) to starting to move the patient from the scene to the helicopter (if intubation in-ambulance, time from entering patient zone until starting to move the patient to the helicopter).
Scene time 2 | While handling the patient case
  Measured from entering patient zone (<3 m) to declaring pilot can switch on helicopter motors.
Ground time | While handling the patient case
  Mesaured from physician leaves helicopter to declaring pilot can switch on helicopter motors.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Gellerfors, Principal Investigator — A PMI, Karolinska University Hospital, Stockholm
Locations (2):
- Sweden (2):
  - HEMS Dalarna, Mora, Dalarna County
  - HEMS VGR, Gothenburg, VästraGötaland

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From 2022

REFERENCES:
- [Derived] Broms J, Gunther M, Svensen C, Kruger A, Rognas L, Gellerfors M. The impact of airway assistants on prehospital endotracheal intubations - a subgroup analysis of data from anaesthesiologist-staffed helicopter critical care teams. Scand J Trauma Resusc Emerg Med. 2025 Nov 25;33(1):194. doi: 10.1186/s13049-025-01515-y. PMID 41291842
- [Derived] Broms J, Linhardt C, Fevang E, Helliksson F, Skallsjo G, Haugland H, Knudsen JS, Bekkevold M, Tvede MF, Brandenstein P, Hansen TM, Kruger A, Rognas L, Lossius HM, Gellerfors M. Prehospital tracheal intubations by anaesthetist-staffed critical care teams: a prospective observational multicentre study. Br J Anaesth. 2023 Dec;131(6):1102-1111. doi: 10.1016/j.bja.2023.09.013. Epub 2023 Oct 14. PMID 37845108